CLINICAL TRIAL: NCT00304850
Title: Efficacy of a Polyamine-free Diet Associated or Not With Ketamine on Early and Late Hyperalgesia After Breast Cancer Surgery
Brief Title: Polyamine-free Diet to Prevent Post Surgery Hyperalgesia
Acronym: PoLyDOL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry of Health, France (Other Government); Insurance CNP foundation (Unknown)
Responsible Party: Jean-Pierre LEROY / Clinical Research and Innovation Director, University Hospital, Bordeaux
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 9258-03; 2002-004
Record Dates: First submitted 2006-03-17; First posted 2006-03-20 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-12

CONDITIONS: Breast Cancer; Surgery
Keywords: polyamines; pain; breast cancer; mastectomy; post operative pain
MeSH Terms: conditions — Breast Neoplasms; Pain; Pain, Postoperative | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- R+ / K+ (Experimental)
  Interventions: Behavioral: polyamine-free diet; Drug: Ketamine or placebo
- R+ / K- (Experimental)
  Interventions: Behavioral: polyamine-free diet; Drug: Ketamine or placebo
- R- / K+ (Experimental)
  Interventions: Drug: Ketamine or placebo
- R- /K- (Placebo Comparator)
  Interventions: Drug: Ketamine or placebo

INTERVENTIONS:
Behavioral: polyamine-free diet — Polyamine-free diet in the 7 days befor surgery
  Arms: R+ / K+; R+ / K-
Drug: Ketamine or placebo — Peroperative and post operative (48h) ketamine injection

SUMMARY:
After surgery, sensitization and hyperexcitability of central nervous system result in acute and long lasting postoperative pain. It has been shown that N-methyl-D-aspartate (NMDA) receptors antagonist (such as ketamine) prevent this adverse neuroplasticity and potentiate analgesic drugs efficacy. Polyamines (putrescine, spermidine, spermine) are essential components of cells functioning and are also known as allosteric modulators of NMDA receptors. In animal studies, polyamine-free diet has confirmed these antinociceptive properties. This research aims at evaluating anti hyperalgesic properties of polyamine-free diet in women operated on breast cancer versus kétamine

DETAILED DESCRIPTION:
This multicentric, single blind study will enrol 160 women (18-75 years old) operated on tumorectomy and adenectomy (T1, T2, T3, N0, N1, M0) for breast cancer. Patients will be randomly assigned in a 2x2 factorial plan : Group 1 = control (n = 40) ; group 2 = ketamine group administered during and 48 hours after a standardized anesthesia (n = 40) ; group 3 = polyamine-free diet, 1 week and 72 hours after surgery (n = 40) ; group 4 : ketamine + polyamine-free diet (n = 40).

The amount of morphine for the 24 first postoperative hours will be compared between each group as well as pain score, allodynia (Von Frey filaments) and hyperalgesia (algometer). Chronic pain occurrence (post-mastectomy pain syndrome) will be evaluated at 3 and 6 months using adequate questionnaire ( analgesic scale). Diet observance will be controlled preoperatively by a dosage of polyamines in circulating red cells blood.

Polyamines deprivation and ketamine ability to reduce postoperative pain will be compared (isobolographic method). Anti-hyperalgesic properties of ketamine have already been demonstrated in urologic, orthopaedic and abdominal surgery. In case of additive or synergistic effect of a polyamine deprivation such a strategic could be helpful to achieve better postoperative rehabilitation in reducing chronic pain after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer (T1, T2, T3, N0, N1, M0)
* Age : 18 - 75
* Asa 1-3
* left or right tumorectomy with complete lymphadenectomy
* left or right complete mastectomy with complete lymphadenectomy
* complete lymphadenectomy within one week following simple tumorectomy
* informed consent signed

Exclusion Criteria:

* inflammatory tumor requiring pre-operative radiotherapy
* previous history of total mastectomy or partial contralateral mastectomy
* chronic inflammatory disease treated by corticoids or NSAI
* chronic analgesic treatment
* anti-arrhythmic or anti-epileptic treatments
* morphinic treatment during the 7 days before surgery
* excessive alcohol consumption or addiction
* ketamine or neomycin contra-indication
* severe cardiovascular disease

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2006-03; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Morphine requirement | for the 24 postoperative hours

SECONDARY OUTCOMES:
Pain intensity for the 4 days (and possibly at 7th day if the patient is still hospitalized) after surgery | 4 days
Allodynia measurements | inclusion, 1, 2, 4 and 7 ddays after surgery
Hyperesthesia measurements | inclusion, 1, 2, 4 and 7 ddays after surgery
Chronic pain incidence | 3 and 6 months
Late allodynia and/or hyperesthesia | 6 months
safety of treatment | Along each patient folow-up

CONTACTS AND LOCATIONS:
Overall Officials: Pierre MAURETTE, Pr, Principal Investigator — DAR 3 -Pellegrin hospital-33076 Bordeaux - France; Genevieve CHENE, Pr, Study Chair — University hospital - 33076 Bordeaux - France
Locations (5):
- France (5):
  - CLCC-Institut Bergonie, service d'anesthésie réanimation, 229 cours de l'Argonne, Bordeaux
  - département d'anesthésie-réanimation 3, hôpital Pellegrin, Bordeaux
  - CLCC Alexis Vautrin, Nancy
  - APHParis Hôpital Pitié Salpétrière - Dépt. d'anesthésie réanimation, Paris
  - CLCC Réné Huguenin de Saint Cloud, Saint-Cloud